CLINICAL TRIAL: NCT02393469
Title: Effects of Pulmonary Rehabilitation on Function Cardiovascular, Respiratory and Functional Capacity of People With Chronic Obstructive Pulmonary Disease in the Municipality of Santa Cruz do Sul - Rio Grande do Sul.
Brief Title: Effects of Pulmonary Rehabilitation on Respiratory, and Cardiovascular Functional Capacity in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Santa Cruz do Sul (Other)
Responsible Party: Principal Investigator, Andrea Lucia Gonçalves da Silva, Doctor, University of Santa Cruz do Sul
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RP_01
Record Dates: First submitted 2014-09-02; First posted 2015-03-19 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status; Self-Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group phase 1 (Placebo Comparator): Two months of education and self-management for COPD where patients know their disease, pathophysiology, treatment, exacerbation of symptoms, and better ways pharmacological treatment education will be conducted through a system of multidisciplinary lessons with professional Physiotherapists, Psychologists, Dieticians, Pharmacists , Physical Education Professionals and Doctors
  Interventions: Other: Education and self-management for COPD
- Group phase 2 (Experimental): Pulmonary rehabilitation for two months: The same patients enter phase 1 phase 2 performing this two months of pulmonary rehabilitation are also included new patients who participate directly in phase 2
  Interventions: Other: pulmonary rehabilitation
- Group phase 3 (Experimental): Pulmonary rehabilitation for ten months: Participate participants of phases 1 + 2 and 2, as well as new participants enter directly in phase 3
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — Exercises breathing exercises are performed on a cycle ergometer for 30 minutes, monitored by 50% of your maximum heart frequency, strengthening exercises for major muscle groups of the upper and lower limbs with charges based on 70% of one repetition maximum, muscle stretching test, and in expiratory pattern
  Arms: Group phase 2; Group phase 3
Other: Education and self-management for COPD — Two months of continuous and self management for COPD where patients know their disease, pathophysiology, treatment, exacerbation of symptoms, and better ways pharmacological treatment education will be conducted through a system of multidisciplinary lessons with professional Physiotherapists, Psychologists, Dieticians, Pharmacists , Physical Education Professionals and Doctors
  Arms: Group phase 1

SUMMARY:
The Chronic Obstructive Pulmonary Disease (COPD) has shown a progressive increase of morbidity and mortality, suggesting that the lung as a single therapeutic target, has not contributed in the past 20 years, significant changes to the natural evolution of the disease. Direct treatment for systemic changes and comorbidities, in fact, the most responsible for high rates of treatment failure could mean a new hope of life for individuals with COPD. This research project characterized as interdisciplinary and multidisciplinary program will be headquartered in Pulmonary Rehabilitation of the Santa Cruz Hospital which has partnerships with local companies . Its main objective will be to analyze cardiorespiratory and functional capacity in COPD patients not rehabilitated and rehabilitated after the period from 02 to 12 months of treatment in a Pulmonary Rehabilitation program in the municipality of Santa Cruz do Sul - Rio Grande do Sul. Will be included in this survey of COPD patients who were referred to a rehabilitation program with a clinical diagnosis of disease. In research activities to assess cardiorespiratory and functional capacity of COPD, pre and post-program (02 and 12 months) are provided for Pulmonary Rehabilitation. The research subjects will also be subjected to physical exercise protocol as recommended by the GOLD (2009), a period of eight weeks, often 2x / week, where their vital signs are measured before, during and after each session. Thus, it is believed that it will be possible to refine the knowledge of mechanisms by which the judicious use of pulmonary rehabilitation can control the progression of COPD.

DETAILED DESCRIPTION:
Selection of project participants

COPD, duly diagnosed with proof of spirometric lung function, who are receiving outpatient care at the Hospital Santa Cruz (HSC) to compose the control group will be selected. For Rehabilitation Pulmonary Group fase 01 (GRP1) and Rehabilitation Pulmonary Group fase 02 (GRP2) will be selected COPD patients who participate in the program Rehabilitation Pulmonary occurring within the HSC, in the municipality of Santa Cruz do Sul - Rio Grande do Sul. The sample size calculation is performed according to the primary endpoint of the study.

All individuals involved in the project have signed a term of informed consent and answer a questionnaire of personal health, containing demographic information, exposure to radiation and drugs, as well as eating habits and consumption of alcohol and cigarettes.

Methodological procedures

The methodological steps of the study will consist of:

1. Selection of subjects according to the criteria of inclusion and exclusion;
2. As an outpatient treatment without Pulmonary Rehabilitation (PR) assess lung volumes, respiratory muscle strength, dyspnea for Medical Research Council (MRC), functional capacity for Functional Independence Measurement (MIF) and Six Minutes Walk Test (6MWT), grip strength, Quality of Life (QoL), body mass index (BMI), and ankle-brachial index (ITB);

4) As a submission to Rehabilitation Pulmonary after 02 months of treatment to assess lung volumes, respiratory muscle strength, MRC, functional capacity (MIF and 6MWT), grip strength, QoL, BMI, and ITB; 5) As a submission in Rehabilitation Pulmonary after 12 months of treatment to assess lung volumes, respiratory muscle strength, MRC, functional capacity (MIF and 6MWT), grip strength, QoL, BMI, and ITB

Techniques and tools for collecting

Lung volumes Lung volumes will be assessed through digital spirometry (EasyOne ®, Model 2001, Zurich, Switzerland). It is a tool to provide a record of several volumes and airflows that an individual is able to mobilize, as the gold standard for assessment of pulmonary functions according to the International Guidelines of the Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2011). Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), forced expiratory flow between 25% and 75% of FVC (FEF 25% -75%), FEV/FVC relationship, (In the present study, the following variables will be evaluated FEV1 / FVC) and peak expiratory flow (PEF) (GONTIJO, 2011). Three measures and the curve that presents the best performance will be compared with the predicted values in the literature and described in percentage of predicted will be realized (Pereira et al., 1992).

Respiratory Muscle Strength (FMR)

The FMR (MIP and MEP) will be evaluated through digital manometer (MDI®, Porto Alegre, Brazil). The MIP will be obtained after the individual expiration to residual volume (RV), the examiner connected with the nose clip and requested inspiration to total lung capacity (TLC). The MEP will be evaluated after the Total Lung Capacity inspiration to the residual volume the mouthpiece (ATS, 2002). For data analysis, will be considered the highest value among the five maneuvers, which did not differ more than 10% of the second highest value in descending order. These values are then compared with those reported in the literature (NEDER et al., 1999) and expressed as percentage of predicted. It is noteworthy that for these measures, the patient will remain in sitting position in the chair or sitting on the bed with an inclination of 45 °.

Functional dyspnea

The MRC (Medical Research Council), which is a British medical institute, developed a scale to graduate dyspnea in patients with COPD. The MRC scale is used for decades and has been adapted into Portuguese and published in published in the II Brazilian Consensus on COPD (2004). Patients were originally categorized into five grades, ranging from 1 ("normal") to 5 ("very dyspneic to leave the house"). The scale focuses primarily on dyspnoea occurring on walks. The MRC scale is widely used in patients with COPD due to its simplicity, ease of use and correlation with quality of life and prognosis.

Functional Capacity

Functional capacity is the independence of an individual to accomplish their mental and physical activities to maintain their basic and instrumental activities.

The Functional Independence Measure (FIM) is an assessment tool for people in the rehabilitation process, part of the Uniform Data System for Medical Rehabilitation (SUDRM) and is widely used and accepted internationally as a measure of functional assessment. Is linked to mobility and functional capacity in which the individual does not require help to perform the same, ie, independence supposed to satisfactory performance of motor and cognitive tasks conditions. The use of the scale focuses on the effective realization of activities independently in daily routine. So lets documenting their sensitivity to functional acquisitions and its correlation with functional levels.

The degree of dependence is classified according to the functional independence measure. This instrument consists of six dimensions: self-care, sphincter control, transfers, locomotion, communication and social cognition. Each item scores from 1 (total dependence) to 7 (complete independence). Obtain minimum total score of 18 and maximum of 126 points that characterize the levels of dependence. Through the individual score will be classified as follows: mild disability (> 80 points), moderate disability (40-80 points) or severe disability (<40).

To perform the 6MWT is the standard protocol used ATS Six-Minute Walk Test (2002). The 6MWT will be held itself, 02 tests, a practice test for educational purposes and another 6MWT, which will be validated for the collected information of the distance walked in six minutes and done. Standard phrases of encouragement will be given by the examiner and if necessary, subjects receive during testing, supplemental oxygen (O2) to maintain a peripheral O2 saturation above 90%.

Dynamometry Manual

Evaluation of peripheral muscle strength by Dynamometry Manual (DM) appears as a simple, objective, low cost alternative and less invasive to measure maximal voluntary handgrip strength and its principle to estimate the function of skeletal muscle. The dynamometer is a device simple to use, and provides fast and direct reading. This test enables indicating health risks related to muscle strength and correlated to other skeletal muscles in the human body, and is considered a good indicator for the overall muscle strength and also to assess physical performance in several clinical situations. Conform the American Society of Hand Therapist (ASHT), for measuring handgrip, patients should be seated comfortably with adducted and neutrally rotated, elbow flexed at 90 °, with arm in neutral pronation-supination and shoulder wrist joint between 0 ° and 30 ° of extension. The procedure should be performed three times in both limbs (right and left) the average of the measurements of each hemibody being calculated separately and given a resting time of 60 seconds between ume measurement and another quoted by.

Quality of Life (QOL)

The questionnaire St. George's Respiratory Questionnaire (SGRQ) which is specific for the assessment of QoL in patients with COPD will be used. This questionnaire consists of 76 items and is divided into 03 domains (symptoms, activity and impact of the disease). For each domain, the items are coded and transformed into a scale of zero (worst QOL) to 100 points (best QoL), according to the standardization of the Manual.

Anthropometric Assessment

The most widely used anthropometric measurements to assess nutritional status are: weight, height, circumferences (arm and waist), arm length and skinfold thicknesses (triceps, biceps, subscapular, suprailiac). Through the combination of these measures is possible to calculate the weight / height, arm muscle circumference and arm fat index relationships.

Anthropometric measurements are easy to perform and relatively sensitive to evaluate adult patients hospitalized in isolation as malnutrition. The body mass index (BMI), expressed as the relationship between body mass in kg and height in m2, is widely used as an indicator of nutritional status for its good correlation with body mass and low correlation with height.

Ankle-Brachial Index (ABI)

The ABI is a noninvasive measurement of peripheral arterial disease is highly predictive of subsequent cardiovascular morbidity and mortality in hypertensive patients. It is the relationship between the (maximum) of the ankle systolic blood pressure (right and left) and the (maximum) arm systolic blood pressure (right and left) with the patient at rest which is taken as a reference the largest value observed among measured the sides. Gauging the (maximum) systolic blood pressure of lower limbs is taken through the ankle being performed using a Doppler Vascular Portable and upper limbs with a sphygmomanometer. It will be noted that the ankle pressure is generally higher, then a ratio of 1 to 1.1 is normal. It is noteworthy that a lower index 0.9 provides strong evidence of peripheral arterial disease, thus the lower the value, the more severe the disease, as this reduction is due to the presence of arterial obstruction in the lower limb. This index is strongly associated with the incidence of strongly related to the individual's functional capacity Arterial Chronic Disease.

Waist-Hip Ratio (WHR)

To obtain the WHR, the waist is measured at the narrowest part of the waist, between the last rib and the iliac crest and hip circumference is taken at the widest area of the hips and the largest protuberance of the buttocks. Then divide the waist measurement by the hip measurement. WHO defines the indices of> 9.0 in men and> 8.5 in women as a crucial relationship to the metabolic syndrome. Studies confirm and cite several other studies that show that WHR is superior to predict all-cause and cardiovascular disease mortality clinical measure. Another Study add that the hip circumference indicates a lower risk of body fat accumulation and thus include it in the waist-hip ratio equation improves the accuracy of the measurement technique.

Lactate analysis

In conjunction with the 6MWT, the measure of capillary lactate could estimate muscle metabolism profile of COPD patients, since his early increase before the physical exertion seems to be associated with changes in muscle metabolism, observable loss of oxidative activity of skeletal muscle . The measurement will be performed after obtaining a drop of capillary blood from the tip of the second finger of the nondominant hand for analysis of lactate at rest and after the 6MWT, the pre-Rehabilitation Pulmonary intervals, 02, and 12 months post-Rehabilitation Pulmonary, (Lct) on the in lactate analyzer Accutrend Plus.

Intervention procedures

The group of patients undergoing Rehabilitation Pulmonary will carry out the intervention protocol as recommended by the GOLD (2009). Will undergo submaximal aerobic training for 30-40 minutes strength training for upper and lower limbs, muscle stretching, nutritional and pharmacological monitoring and continuing education sessions, twice a week. Such measures will be carried out under the Hospital Santa Cruz, Santa Cruz do Sul - Rio Grande do Sul.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with a clinical diagnosis

Exclusion Criteria:

* Motor sequelae of stroke, patients undergoing treatment for infectious diseases, musculoskeletal disorders that impede ambulation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Functional capacity in COPD patients | Will initially be evaluated after ten months.

SECONDARY OUTCOMES:
Ankle brachial index | Will be assessed after the admission of patients to pulmonary rehabilitation program. will be held after admission, subsequently after two and ten months
  The ankle brachial index is a noninvasive test used to evaluate the arterial blood flow in the lower limbs, is highly sensitive for the detection of peripheral arterial disease
Window in ischemic lower limbs | will be evaluated after functional testing submaximal. will be held after admission, subsequently after two and ten months
  Along with Ankle-Brachial Index, after the six-minute walk test will be rated at 2, 4 and 6 minutes after the test which may be obtained, or not, an ischemic curve in COPD patients
walk test six minutes | will be conducted to evaluate rates of ischemic window by ankle brachial index, will be held after admission, subsequently after two and ten months
  The test of six-minute walk test is a functional capacity and secondarily submaximal cardiovascular function, where the individual will need to walk for six minutes at maximum speed, without running.
heart rate variability | will be held Durantes three tests: Shuttle Walk Test, test and six-minute walk incremental protocol in cycle rgometer. will be held after admission, subsequently after two and ten months
  The heart rate variability assesses the R-R curves of the electrocardiographic tracing of the heart using a heart rate monitor and is currently used to evaluate the sympathetic-vagal activity of the heart. In our study we use in all tests with patients (Astrand Protocol treadmill, Shuttle Walk Test and the Six Minute Walk Test)
Shuttle Walk Test | Will be conducted to evaluate the functional capacity of the study participants. will be held after admission, subsequently after two and ten months
Incremental protocol in cycle ergometer (Astrand Treadmill test) | will be held in conjunction with analysis of the lactate curve to assess the ability of resistance to fatigue of the participants, will be held after admission, subsequently after two and ten months
  The incremental Astrand Treadmill Test, is an incremental test on a cycle ergometer vertical predicts that the maximum capacity of an individual's body to transport and metabolize oxygen during incremental exercise. Together with this test will be evaluated index blood lactate every 3 minutes of testing.
assessment of lung function | will be held after the admission of patients to the project, will be held after admission, subsequently after two and ten months
  Lung function at digital spirometry assesses lung volumes through the forced vital capacity maneuver. Allows detecting obstructive, restrictive or mixed disorders.
assessment of respiratory muscle strength | will be held after admission, subsequently after two and ten months
  Respiratory muscle strength will be assessed through maximal respiratory pressures test and helps assess maximal expiratory and inspiratory force through the pressures generated by the patient. This test evaluates jointly the inspiratory muscles, and likewise the expiratory muscles.
assessment of handgrip strength | will be held after admission, subsequently after two and ten months
  The grip strength will be assessed by hydraulic handgrip dynamometer. It is a test that evaluates the strength of the handshake individual and quantifies overall muscle strength.
assessment of quality of life | will be held after admission, subsequently after two and ten months
  The quality of life will be assessed through the questionnaire Saint George's Respiratory Questionnaire. It is created and validated a questionnaire focused for patients with respiratory diseases.
assessment of the economic and social level | will be evaluated only once
  The socioeconomic level of the individuals will be assessed by the Brazilian Association of Research Companies survey. It is a questionnaire created in Brazil to quantify the economic track of the Brazilian population specifically.
classification of patients as BODE index | Will be assessed at baseline (start of pulmonary rehabilitation) and after 10 months (final evaluation)
  The BODE index is an index that assesses the health status of patients with COPD. It consists of four items (B - measured by body mass index or "body mass in-dex" (weight / height); O - obstruction as measured by FEV1 (forced expiratory volume in one second); D - measured by degree of dyspnea; E - exercise, assessed by using the 6-minute walk)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Gonçalves da Silva, Doctor, Principal Investigator — University of Santa Cruz do Sul; Dulciane N Paiva, Doctor, Study Director — University of Santa Cruz do Sul; Dannuey M Cardoso, Ms, Study Chair — University of Santa Cruz do Sul; Diogo F Bordin, Academic, Study Chair — University of Santa Cruz do Sul; Ricardo Gass, Academic, Study Chair — University of Santa Cruz do Sul; Cássia L Goulart, Academic, Study Chair — University of Santa Cruz do Sul; Natacha Angélica M da Fonseca, Academic, Study Chair — University of Santa Cruz do Sul; Camila da C Niedermeyer, Academic, Study Chair — University of Santa Cruz do Sul; Lisiane L Carvalho, Msc, Study Chair — University of Santa Cruz do Sul
Locations (1):
- Universidade de Santa Cruz do Sul, Santa Cruz do Sul, Rio Grande do Sul, Brazil